CLINICAL TRIAL: NCT04905641
Title: The Feasibility of Bilateral Intermediate Cervical Plexus Block for Thyroidectomy/Parathyroidectomy Under Moderate Sedation; Retrospective Study
Brief Title: The Feasibility of Bilateral Intermediate Cervical Plexus Block for Thyroidectomy/Parathyroidectomy
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Suwimon Tangwiwat, Department of Anesthesiology, Mahidol University
Other Study IDs: Si 081/2018
Record Dates: First submitted 2021-05-26; First posted 2021-05-27 (Actual); Last update posted 2021-06-01 (Actual); Status verified 2021-05

CONDITIONS: Parathyroid Adenoma; Thyroid Nodule
Keywords: intermediate cervical plexus block
MeSH Terms: conditions — Parathyroid Neoplasms; Thyroid Nodule

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Bilateral intermediate cervical plexus block — Bilateral intermediate cervical plexus block was performed under ultrasound guidance.

SUMMARY:
The aim of this study was evaluated the feasibility of bilateral intermediate cervical plexus blockade to be anesthesia for simple thyroid/parathyroid surgery.

DETAILED DESCRIPTION:
Bilateral intermediate cervical plexus blocks have been reported for thyroid/parathyroid surgery. This technique combined with intravenous sedation has used with safety in patients undergoing simple thyroid or parathyroid surgery. Simple surgery is defined as the thyroid conditions are not cancer, redo or substernal goiter.

ELIGIBILITY:
Inclusion Criteria:

* patient underwent thyroid/parathyroid surgery under nerve blocks and sedation

Exclusion Criteria:

* incomplete opioid consumption or pain score record.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: bilateral intermediate cervical plexus block for thyroid nodule or parathyroid adenoma
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2016-03-10 (Actual); Primary Completion 2017-05-25 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Conversion to general anesthesia | during operation
  inability to operate under nerve block and sedation

SECONDARY OUTCOMES:
opioid usage | intraoperative
  fentanyl consumption
dypnea | intraoperative
  phrenic nerve paralysis
pain score within 24 hours | within 24 hours postoperative
  numerical rating score
complications | intraoperative
  local anesthetic systemic toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Suwimon Tangwiwat, MD, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Arora N, Dhar P, Fahey TJ 3rd. Seminars: local and regional anesthesia for thyroid surgery. J Surg Oncol. 2006 Dec 15;94(8):708-13. doi: 10.1002/jso.20694. PMID 17131394
- [Result] Spanknebel K, Chabot JA, DiGiorgi M, Cheung K, Lee S, Allendorf J, Logerfo P. Thyroidectomy using local anesthesia: a report of 1,025 cases over 16 years. J Am Coll Surg. 2005 Sep;201(3):375-85. doi: 10.1016/j.jamcollsurg.2005.04.034. PMID 16125070
- [Result] Yerzingatsian KL. Thyroidectomy under local analgesia: the anatomical basis of cervical blocks. Ann R Coll Surg Engl. 1989 Jul;71(4):207-10. PMID 2774445
- [Result] Plunkett AR, Shields C, Stojadinovic A, Buckenmaier CC. Awake thyroidectomy under local anesthesia and dexmedetomidine infusion. Mil Med. 2009 Jan;174(1):100-2. doi: 10.7205/milmed-d-01-2908. PMID 19216305
- [Result] Egan RJ, Hopkins JC, Beamish AJ, Shah R, Edwards AG, Morgan JD. Randomized clinical trial of intraoperative superficial cervical plexus block versus incisional local anaesthesia in thyroid and parathyroid surgery. Br J Surg. 2013 Dec;100(13):1732-8. doi: 10.1002/bjs.9292. PMID 24227357
- [Result] Jung KJ, Park JY, Hwang DW, Kim JH, Kim JH. Ultrasonographic diaphragmatic motion analysis and its correlation with pulmonary function in hemiplegic stroke patients. Ann Rehabil Med. 2014 Feb;38(1):29-37. doi: 10.5535/arm.2014.38.1.29. Epub 2014 Feb 25. PMID 24639923
- [Result] Boussuges A, Gole Y, Blanc P. Diaphragmatic motion studied by m-mode ultrasonography: methods, reproducibility, and normal values. Chest. 2009 Feb;135(2):391-400. doi: 10.1378/chest.08-1541. Epub 2008 Nov 18. PMID 19017880